CLINICAL TRIAL: NCT00531804
Title: A Multi-center, Multiple-ascending Dose, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO4909832 Following Intravenous Infusion in AD Patients
Brief Title: A Multiple Ascending Dose Study of R1450 in Patients With Alzheimer Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN19866
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — gantenerumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: gantenerumab

INTERVENTIONS:
Drug: gantenerumab — Administered iv at escalating doses (7 cohorts)

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of R1450 in patients with mild to moderate Alzheimer Disease. Patients will be randomized to receive either R1450 or placebo by intravenous infusion for a total of 7 doses. The starting dose will be escalated in subsequent cohorts of patients in an adaptive manner, after a satisfactory assessment of safety, tolerability and pharmacokinetics of the previous dose. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 50-90 years of age;
* diagnosis of probable Alzheimer Disease, with symptoms >=1 year prior to screening;
* meets DSM-IV criteria for Alzheimer-type dementia;
* stabilised on approved medications for treatment of Alzheimer Disease for >=4 months prior to baseline.

Exclusion Criteria:

* active major depressive disorder, or a history of bipolar disorder;
* history of schizophrenia;
* concurrent participation in a non-pharmacological trial with a key objective of improving cognition;
* prior randomisation in any R1450 trial.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
AEs, laboratory parameters, vital signs. | Throughout study
Pharmacokinetic parameters of R1450 in plasma | Throughout study

SECONDARY OUTCOMES:
CSF biomarkers, clinical efficacy parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Copenhagen, Denmark
- Ramat Gan, Israel
- Amsterdam, Netherlands
- Sweden (2):
  - Malmo
  - Stockholm
- United Kingdom (4):
  - Blackpool
  - Glasgow
  - Southampton
  - Swindon